CLINICAL TRIAL: NCT03432819
Title: A Pilot Intervention to Improve Coping With Discrimination and Adherence Among HIV-Positive Latino MSM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RAND (Other)
Collaborators: Bienestar Human Services, Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R34MH113413 (NIH)
Record Dates: First submitted 2018-01-31; First posted 2018-02-14 (Actual); Results first posted 2021-02-25 (Actual); Last update posted 2023-03-29 (Actual); Status verified 2023-03

CONDITIONS: HIV
Keywords: Latino, men who have sex with men
MeSH Terms: conditions — Homosexuality

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Siempre Seguiré (Experimental): We will conduct a small randomized controlled trial (RCT), testing study protocols and materials, the acceptability of randomization, and overall program feasibility. The pilot will help to identify logistical considerations; assess whether the program is acceptable and understandable LMSM; and collect initial data on how successfully the program motivates change in coping and adherence. It will allow us to estimate expected attrition and response rates, and to perform preliminary power analyses in preparation for a fully powered RCT.
  Interventions: Behavioral: Siempre Seguiré
- Control (No Intervention): Control participants will not be randomized to receive the intervention and will receive standard of care during the intervention period. We will offer the program to any interested control participants shortly after the 6-month follow-up surveys are completed.

INTERVENTIONS:
Behavioral: Siempre Seguiré — A culturally congruent CBT group intervention for HIV-positive LMSM, to include strategies for ART adherence and retention in HIV care.
  Arms: Siempre Seguiré

SUMMARY:
R34-funded study to pilot test an intervention to improve coping with discrimination and adherence among Latino men who have sex with men (MSM) living with HIV. The proposed research aims to modify and refine Siempre Seguiré, a culturally congruent cognitive behavior therapy group intervention for HIV-positive Latino men who have sex with men (LMSM), to include strategies for ART adherence and retention in HIV care; and to conduct a small randomized pilot of Siempre Seguiré to examine feasibility and acceptability, as well as to explore preliminary effects on coping responses to discrimination and antiretroviral treatment adherence among LMSM living with HIV.

DETAILED DESCRIPTION:
HIV-related disparities in diagnosis and disease outcomes persist among Latinos, and Latinos living with HIV show a lower percentage of viral suppression compared to the general HIV-positive population. A growing body of work suggests that stigma and discrimination contribute to health disparities, especially among people living with HIV, who may experience discrimination due to multiple stigmatized identities related to HIV-serostatus, race/ethnicity, and sexual orientation. Internalized stigma and discrimination may lead to health-related disparities by increasing detrimental physiological stress responses, resulting in maladaptive coping and poor health behaviors, including non-adherence to treatment. Moreover, the chronic stress of discrimination may weaken immune function, leading to worse HIV outcomes, including increased HIV viral load. The proposed research will integrate adherence skills-building strategies into a recently developed intervention, Siempre Seguiré, an 8-session group cognitive behavioral therapy (CBT) intervention for HIV-positive Latino men who have sex with men (LMSM) that aims to improve adaptive coping responses to discrimination. The specific aims are: (1) To modify and refine Siempre Seguiré, a newly developed culturally congruent CBT group intervention for HIV-positive LMSM, to include strategies for antiretroviral treatment adherence and retention in HIV care; and (2) To conduct a small randomized pilot of Siempre Seguiré to examine feasibility and acceptability, as well as to explore preliminary effects on: (a) coping responses to discrimination; and (b) antiretroviral treatment adherence, viral load suppression, and HIV care retention, among LMSM living with HIV. In Phase 1, HIV treatment adherence intervention experts and key stakeholders, including a community advisory board, will help to refine our pilot intervention as needed and update our manual to integrate information and skills building regarding HIV treatment adherence and retention in care. In Phase 2, a small randomized controlled trial of 80 participants (40 intervention participants divided evenly over 4 intervention groups vs. 40 wait-list control participants) will be conducted. Participants will complete surveys at baseline, and 4- and 6-months post-baseline to assess coping and HIV care processes and outcomes. Adherence will be electronically monitored, and viral load will be collected from medical providers at baseline and at 6-month follow-up. Intervention group sessions will take place once per week for 8 weeks. Sessions will take place in a private room at Bienestar (a Latino-serving AIDS service organization in LAC) and will last approximately 90 minutes. We hypothesize that the intervention will improve coping responses to discrimination and HIV treatment adherence.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years-old or older, HIV-positive, biologically male at birth and continue to identify as male, identify as Latino, report having sex with men in the past 12 months, and prescribed ART.

Exclusion Criteria:

* Being unwilling or unable to provide informed consent; having mental health problems that require immediate treatment (e.g., psychotic symptoms) or a diagnosed mental disorder that would limit ability to participate (e.g., dementia); and cognitive impairments that result in limited ability to provide informed consent.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Biologically male at birth and continue to identify as male
Enrollment: 82 (Actual)
Dates: Start 2018-03-27 (Actual); Primary Completion 2019-09-12 (Actual); Study Completion 2019-09-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Laura Bogart, PhD, Principal Investigator — RAND
Locations (1):
- Bienestar Human Services, Inc., Los Angeles, California, United States

REFERENCES:
- [Derived] Barreras JL, Bogart LM, MacCarthy S, Klein DJ, Pantalone DW. Discrimination and adherence in a cross-sectional study of Latino sexual minority men with HIV: Coping with discrimination as a mediator and coping self-efficacy as a moderator. J Behav Med. 2023 Dec;46(6):1057-1067. doi: 10.1007/s10865-023-00426-6. Epub 2023 Jul 1. PMID 37392342
- [Derived] Bogart LM, Barreras JL, Gonzalez A, Klein DJ, Marsh T, Agniel D, Pantalone DW. Pilot Randomized Controlled Trial of an Intervention to Improve Coping with Intersectional Stigma and Medication Adherence Among HIV-Positive Latinx Sexual Minority Men. AIDS Behav. 2021 Jun;25(6):1647-1660. doi: 10.1007/s10461-020-03081-z. Epub 2020 Nov 24. PMID 33231847

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Between completing the baseline survey and being randomized 5 participants were lost to follow up and 1 withdrew due to issues related to homelessness.
Groups:
- Siempre Seguiré: We will conduct a small RCT, testing study protocols and materials, the acceptability of randomization, and overall program feasibility. The pilot will help to identify logistical considerations; assess whether the program is acceptable and understandable LMSM; and collect initial data on how successfully the program motivates change in coping and adherence. It will allow us to estimate expected attrition and response rates, and to perform preliminary power analyses in preparation for a fully powered RCT.
  Siempre Seguiré: A culturally congruent CBT group intervention for HIV-positive LMSM, to include strategies for ART adherence and retention in HIV care.
Period: Overall Study
Arm/Group | Siempre Seguiré | Control
Started | 38 | 38
Completed | 31 | 33
Not Completed | 7 | 5
Not completed — Lost to Follow-up | 2 | 2
Not completed — Withdrawal by Subject | 5 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Siempre Seguiré | Control | Total
Number analyzed (Participants) | 38 | 38 | 76
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.4 (12.9) | 53.5 (13.1) | 52.9 (12.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 38 | 38 | 76
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 38 | 38 | 76
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
ART Adherence [Mean (Standard Deviation); unit: % of doses taken, past month] — Population: The baseline analysis population includes only the 66 participants who completed the baseline survey as well as at least one follow-up survey. Of the 76 participants who completed a baseline survey and were randomized, 63 (98.4%) responded to both follow-ups, another 2 responded only to the 4-month FUP, and another 1 responded only to the 7-month FUP, for a total of 66 who responded to at least one FUP (86.8%).
  % of doses taken, past month
    Self-report: number analyzed (Participants) | 32 | 34 | 66
    Self-report | 94.61 (6.62) | 91.08 (8.97) | 92.9 (8.0)
    MEMS: number analyzed (Participants) | 32 | 34 | 66
    MEMS | 89.2 (17.4) | 82.3 (23.5) | 85.9 (20.7)
Coping with discrimination [Mean (Standard Deviation); unit: units on a scale] — We adapted Brief COPE and R-COPE and asked participants how much they responded in a certain way when faced with discrimination. Responses were 1 = I haven't been doing this at all to 4 = I've been doing this a lot. Functional coping included 16 Brief COPE items, e.g., active coping, and three additional items, e.g., avoid certain situations. Dysfunctional coping included 12 Brief COPE items, e.g., denial. Two R-COPE sub scales were created to assess positive religious coping, e.g., secure relationships with a divine force, and negative religious coping, e.g., underlying spiritual tensions. Population: The baseline analysis population includes only the 66 participants who completed the baseline survey as well as at least one follow-up survey. Of the 76 participants who completed a baseline survey and were randomized, 63 (98.4%) responded to both follow-ups, another 2 responded only to the 4-month FUP, and another 1 responded only to the 7-month FUP, for a total of 66 who responded to at least one FUP (86.8%).
  units on a scale
    Functional coping (16 Brief COPE items, plus three additional items): number analyzed (Participants) | 32 | 34 | 66
    Functional coping (16 Brief COPE items, plus three additional items) | 2.74 (0.45) | 2.78 (0.48) | 2.76 (0.49)
    Dysfunctional co[ping (12 Brief COPE items): number analyzed (Participants) | 32 | 34 | 66
    Dysfunctional co[ping (12 Brief COPE items) | 2.09 (0.36) | 2.14 (0.44) | 2.12 (0.41)
    Positive religious coping (R-COPE subscale): number analyzed (Participants) | 32 | 34 | 66
    Positive religious coping (R-COPE subscale) | 1.86 (0.66) | 2.14 (0.62) | 2.00 (0.65)
    Negative religious coping (R-COPE subscale): number analyzed (Participants) | 32 | 34 | 66
    Negative religious coping (R-COPE subscale) | 0.44 (0.48) | 0.25 (0.35) | 0.34 (0.42)
Medical mistrust [Mean (Standard Deviation); unit: units on a scale] — General medical mistrust was measured with the Mistrust of Healthcare Scale. HIV-specific medical mistrust was measured with the HIV Conspiracy Beliefs Scale. Response options for both were: 1 = Strongly Disagree to 5 = Strongly Agree. Population: The baseline analysis population includes only the 66 participants who completed the baseline survey as well as at least one follow-up survey. Of the 76 participants who completed a baseline survey and were randomized, 63 (98.4%) responded to both follow-ups, another 2 responded only to the 4-month FUP, and another 1 responded only to the 7-month FUP, for a total of 66 who responded to at least one FUP (86.8%).
  units on a scale
    General (Mistrust of Healthcare Scale): number analyzed (Participants) | 32 | 34 | 66
    General (Mistrust of Healthcare Scale) | 2.53 (1.10) | 2.90 (0.96) | 2.71 (1.03)
    HIV Conspiracy Beliefs (HIV Conspiracy Beliefs Scale): number analyzed (Participants) | 32 | 34 | 66
    HIV Conspiracy Beliefs (HIV Conspiracy Beliefs Scale) | 2.33 (1.06) | 2.30 (0.94) | 2.32 (0.99)
Internalized stigma (HIV) [Mean (Standard Deviation); unit: units on a scale] — Internalized HIV stigma was assessed with the Internalized AIDS-Related Stigma Scale . Internalized sexual minority stigma was assessed with the Internalized-Homophobia Scale-Revised. Response options for both were 1 = Strongly Disagree to 5 = Strongly Agree. Population: The baseline analysis population includes only the 66 participants who completed the baseline survey as well as at least one follow-up survey. Of the 76 participants who completed a baseline survey and were randomized, 63 (98.4%) responded to both follow-ups, another 2 responded only to the 4-month FUP, and another 1 responded only to the 7-month FUP, for a total of 66 who responded to at least one FUP (86.8%).
  units on a scale
    Internalized sexual minority stigma: number analyzed (Participants) | 32 | 34 | 66
    Internalized sexual minority stigma | 1.70 (0.96) | 1.84 (0.84) | 1.77 (0.90)
    Internalized HIV stigma: number analyzed (Participants) | 32 | 34 | 66
    Internalized HIV stigma | 2.76 (1.20) | 2.54 (0.88) | 2.65 (1.04)

OUTCOME MEASURES:

1. Primary Outcome: Continuous Adherence (MEMS)
Description: Percentage of doses taken, of those prescribed, from electronic monitoring
Time Frame: 4-5 and 6-7 months post-baseline
Population: Follow-ups were combined and analyzed together, so the analysis population includes only the 66 participants who completed the baseline survey as well as at least one follow-up survey.
Measure: Mean (Standard Deviation); unit: % of doses taken, past month
Arm/Group | Siempre Seguiré | Control
Number analyzed (Participants) | 32 | 34
% of doses taken, past month
  MEMS, 4-5 months post-baseline | 86.7 (16.0) | 79.0 (23.0)
  MEMS, 6-7 months post baseline | 85.5 (19.8) | 79.7 (19.9)
Statistical Analysis 1: Comparison: Siempre Seguiré vs Control; Test type: Superiority — Using an intent-to-treat approach, intervention efficacy was tested with a hierarchical linear repeated-measures regressions where responses came from either follow-up, and MEMS adherence from 5, 6, or 7 month measurements. Predictors were an indicator for study arm, baseline value, follow-up time-point, and covariates. Standard errors were adjusted for clustering at the individual-level (ultimate clustering methods). Covariates were socio-demographics associated with the outcome at p>.05; p = 0.06, Regression, Linear; Mean Difference (Net) = 9.24, 95% CI 2-sided [-0.55 to 19.03]

2. Primary Outcome: Continuous Adherence (Self-report)
Description: Percentage of doses taken, of those prescribed, self-report
Time Frame: 4 and 7 months post-baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: % of doses taken, past month
Arm/Group | Siempre Seguiré | Control
Number analyzed (Participants) | 32 | 34
% of doses taken, past month
  4-month follow-up | 97.48 (5.42) | 94.57 (6.56)
  7-month follow-up | 99.17 (1.51) | 92.91 (16.78)
Statistical Analysis 1: Comparison: Siempre Seguiré vs Control; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.02, Regression, Linear; Mean Difference (Final Values) = 4.50, 95% CI 2-sided [0.70 to 8.30]

3. Secondary Outcome: Functional Coping Strategies
Description: Functional coping strategies as measured by 16 Brief COPE items on active coping, acceptance, social support, positive reframing, planning, humor, and religion, and three additional functional coping items based on prior qualitative research on coping in communities of color ("I tell myself that other people are ignorant"; "I avoid certain situations or people so that I am not discriminated against in the future"; and "I change the way that I dress or talk so that I am not discriminated against in the future"). Responses were 1 = I haven't been doing this at all, 2 = I've been doing this a little bit, 3 = I've been doing this a medium amount, and 4 = I've been doing this a lot in response to discrimination
Time Frame: 4 and 7 months post-baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Siempre Seguiré | Control
Number analyzed (Participants) | 32 | 34
units on a scale
  4-month follow-up | 2.75 (0.43) | 2.68 (0.36)
  7-month follow-up | 2.82 (0.44) | 2.74 (0.45)
Statistical Analysis 1: Comparison: Siempre Seguiré vs Control; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.39, Regression, Linear; Mean Difference (Final Values) = 0.08, 95% CI 2-sided [-0.10 to 0.26]

4. Secondary Outcome: Positive Religious Coping Strategies
Description: Positive religious coping strategies as measured by an R-COPE sub-scale to assess secure relationships with a divine force/spiritual connectedness. Responses were 1 = I haven't been doing this at all, 2 = I've been doing this a little bit, 3 = I've been doing this a medium amount, and 4 = I've been doing this a lot in response to discrimination
Time Frame: 4 and 7 months post-baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Siempre Seguiré | Control
Number analyzed (Participants) | 32 | 34
units on a scale
  4 months post-baseline | 1.84 (0.85) | 2.08 (0.65)
  7 months post-baseline | 1.72 (0.84) | 2.08 (0.65)
Statistical Analysis 1: Comparison: Siempre Seguiré vs Control; Using an intent-to-treat approach, intervention efficacy was tested with a hierarchical linear repeated-measures regressions where responses came from either follow-up, and MEMS adherence from 5, 6, or 7 month measurements. Predictors were an indicator for study arm, baseline value, follow-up time-point, and covariates. Standard errors were adjusted for clustering at the individual-level (ultimate clustering methods). Covariates were socio-demographics associated with the outcome at p>.05; Test type: Superiority; p = 0.54, Regression, Linear; Median Difference (Final Values) = -0.09, 95% CI 2-sided [-0.37 to 0.20]

5. Secondary Outcome: Dysfunctional Coping Strategies
Description: Dysfunctional/ineffective coping strategies dysfunctional/ineffective as measured by 12 Brief COPE items on denial, substance use, behavioral disengagement, venting, self-blame, and self-distraction. Responses were 1 = I haven't been doing this at all, 2 = I've been doing this a little bit, 3 = I've been doing this a medium amount, and 4 = I've been doing this a lot in response to discrimination
Time Frame: 4 and 7 months post-baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Siempre Seguiré | Control
Number analyzed (Participants) | 32 | 34
units on a scale
  4-month follow-up | 2.05 (0.33) | 2.09 (0.41)
  7-month follow-up | 2.06 (0.38) | 2.09 (0.54)
Statistical Analysis 1: Comparison: Siempre Seguiré vs Control; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p = 0.81, Regression, Linear; Median Difference (Final Values) = -0.02, 95% CI 2-sided [-0.18 to 0.14]

6. Secondary Outcome: Negative Religious Coping Strategies
Description: Negative religious coping strategies as measured by an R-COPE sub-scale to assess underlying spiritual tensions/internal struggles. Responses were 1 = I haven't been doing this at all, 2 = I've been doing this a little bit, 3 = I've been doing this a medium amount, and 4 = I've been doing this a lot in response to discrimination
Time Frame: 4 and 7 months post-baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Siempre Seguiré | Control
Number analyzed (Participants) | 32 | 34
units on a scale
  4 months post-baseline | 0.17 (0.24) | 0.34 (0.52)
  7 months post-baseline | 0.22 (0.40) | 0.30 (0.48)
Statistical Analysis 1: Comparison: Siempre Seguiré vs Control; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p = 0.06, Regression, Linear; Median Difference (Final Values) = -0.18, 95% CI 2-sided [-0.37 to 0.01]

7. Secondary Outcome: Medical Mistrust (General)
Description: General medical mistrust was measured with the Mistrust of Healthcare Scale. Response options were 1 = Strongly Disagree to 5 = Strongly Agree.
Time Frame: 4 and 7 months post-baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Siempre Seguiré | Control
Number analyzed (Participants) | 32 | 34
units on a scale
  4 months post-baseline | 2.34 (0.94) | 2.78 (0.96)
  7 months post-baseline | 2.28 (1.20) | 2.88 (1.08)
Statistical Analysis 1: Comparison: Siempre Seguiré vs Control; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p = 0.16, Regression, Linear; Mean Difference (Final Values) = -0.33, 95% CI 2-sided [-0.78 to 0.13]

8. Secondary Outcome: Medical Mistrust (HIV Conspiracy Beliefs)
Description: HIV-specific medical mistrust was measured with the HIV Conspiracy Beliefs Scale. Response options were 1 = Strongly Disagree to 5 = Strongly Agree.
Time Frame: 4 and 7 months post-baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Siempre Seguiré | Control
Number analyzed (Participants) | 32 | 34
units on a scale
  4 months post-baseline | 1.81 (0.86) | 2.26 (0.90)
  7 months post-baseline | 1.90 (1.03) | 2.40 (0.90)
Statistical Analysis 1: Comparison: Siempre Seguiré vs Control; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p = 0.02, Regression, Linear; Mean Difference (Final Values) = -0.47, 95% CI 2-sided [-0.84 to -0.09]

9. Secondary Outcome: Internalized Stigma (Sexual Orientation)
Description: Internalized sexual minority stigma was assessed with the Internalized-Homophobia Scale-Revised. Response options were 1 = Strongly Disagree to 5 = Strongly Agree.
Time Frame: 4 and 7 months post-baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Siempre Seguiré | Control
Number analyzed (Participants) | 32 | 34
units on a scale
  4 months post-baseline | 1.53 (0.79) | 1.59 (0.69)
  7 months post-baseline | 1.68 (1.06) | 1.59 (0.85)
Statistical Analysis 1: Comparison: Siempre Seguiré vs Control; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p = 0.71, Regression, Linear; Mean Difference (Final Values) = -0.08, 95% CI 2-sided [-0.32 to 0.47]

10. Secondary Outcome: Internalized Stigma (HIV)
Description: Internalized HIV stigma was assessed with the Internalized AIDS-Related Stigma Scale. Response options were 1 = Strongly Disagree to 5 = Strongly Agree.
Time Frame: 4 and 7 months post-baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Siempre Seguiré | Control
Number analyzed (Participants) | 32 | 34
units on a scale
  4 months post-baseline | 2.38 (0.93) | 2.38 (0.98)
  7 months post-baseline | 2.14 (0.90) | 2.65 (1.17)
Statistical Analysis 1: Comparison: Siempre Seguiré vs Control; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p = 0.10, Regression, Linear; Mean Difference (Final Values) = -0.34, 95% CI 2-sided [-0.73 to 0.06]

ADVERSE EVENTS:
Time Frame: 7 months
Arm/Group | Siempre Seguiré | Control
All-Cause Mortality (participants affected / at risk) | 0/38 | 0/38
Serious Adverse Events (participants affected / at risk) | 0/38 | 0/38
Other Adverse Events (participants affected / at risk) | 0/38 | 0/38

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-02-01): https://cdn.clinicaltrials.gov/large-docs/19/NCT03432819/Prot_SAP_001.pdf